CLINICAL TRIAL: NCT05460897
Title: Health Behaviour Change in Brazilians - Effectiveness of a Pan-Canadian English-language Program, Translated Into Brazilian Portuguese, to Increase Healthy Behaviours
Brief Title: Health Behaviour Change in Brazilians
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Darren Warburton, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H17-03564
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Physical Inactivity; Eating Behavior; Smoking
MeSH Terms: conditions — Sedentary Behavior; Feeding Behavior; Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): 12-week intervention consisting of educational sessions and health behaviour change techniques
  Interventions: Behavioral: Health behaviour change
- Waitlist control group (No Intervention): After the first 12 weeks, this group will receive the same intervention as the experimental group

INTERVENTIONS:
Behavioral: Health behaviour change — weekly sessions addressing strategies to tackle behavioural risk factors for chronic disease
  Arms: Experimental

SUMMARY:
Chronic diseases are the leading health problem in Brazil and Canada. Such diseases share common risk factors in common, such as physical inactivity, poor diet, and smoking. This context requires a comprehensive approach to change these behavioural risk factors, aiming at the promotion of healthy lifestyles and the prevention of diseases. Although Brazil and Canada have significant differences, particularly in terms of socioeconomic factors, some similarities in the health domain allow both countries to mutually benefit from an exchange of knowledge. For instance, the newest version of Canada's dietary guidelines has incorporated several aspects presented in the pioneering evidence-based dietary guidelines for the Brazilian population, launched in 2014. Similarly, Brazil can greatly benefit if the country follows the Canadian lead in prioritizing investment in physical activity initiatives. The present project aims to verify the effectiveness of a Canadian program to change health behaviours, specifically physical inactivity, poor diet, and smoking, adapted for Brazilians. The project consists of a 12-week randomized controlled trial, based on education and behaviour change techniques focusing on physical activity, healthy eating habits, and smoking cessation. Pre-, post, and 3-month follow-up health and fitness assessments will evaluate respectively the initial condition of the participants, eventual changes and if the changes persist.

ELIGIBILITY:
Inclusion Criteria:

Brazilians who speak Brazilian Portuguese fluently, and present at least one of the following risk factors:

* physical inactivity (<150 min of MVPA per week)
* unhealthy diet (consumption of fewer than five fruits/vegetables per day)
* smoking (any amount of personal tobacco use)

Exclusion Criteria:

* unstable clinical conditions
* inability to participate fully in the program due to mental or physical limitations
* concurrently participation in other studies of intensive health behaviour modification

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Physical activity | 12 weeks
  change in the proportion of participants engaging in ≥ 150 min moderate to vigorous physical activity (MVPA) per week

CONTACTS AND LOCATIONS:
Overall Officials: Darren Warburton, PhD, Principal Investigator — Professor
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada